CLINICAL TRIAL: NCT00097058
Title: Estrogen Use in Protection From Cognitive Decline
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Natalie Rasgon, Principal Investigator, Stanford University
Other Study IDs: IA0063; R01AG022008 (NIH); SPO #29004; Grant #R01 AG022008; NCT00238589 (obsolete NCT alias)
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Aging; Menopause
Keywords: Aging; Menopause; Estrogen Replacement Therapy; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood serum urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Continue current hormone therapy
- 2: Taper off hormone therapy

SUMMARY:
This study is designed to assess the effects of estrogen therapy among postmenopausal women at risk for cognitive decline.

DETAILED DESCRIPTION:
A total of 71 postmenopausal women ages 50-65 on estrogen therapy will be randomized to continue or discontinue use of estrogen and will be followed for two years.

Participants will undergo PET and MRI scans and neuropsychological assessments initially and at the end of the two-year follow-up period. These procedures will allow us to evaluate brain metabolism and cognitive performance at baseline and two years following continuation or discontinuation of estrogen therapy.

We hypothesize that women who discontinue estrogen will show more evidence of decline than those who continue estrogen. This project will expand current knowledge of effects of estrogen by 1) determining whether estrogen use among postmenopausal women at risk for cognitive decline is protective of brain metabolism, 2) identifying early predictors for cognitive decline, and 3) developing guidelines for estrogen use in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 45 and 65
* Currently on hormone replacement
* One year or more post complete cessation of menses
* Willing to sign the Human Subject Protection Consent form prior to enrollment in the study
* Willing to be randomized to continue or discontinue estrogen therapy
* Adequately visually and auditorially acute to allow neuropsychological testing
* Beyond 8 years of educational achievement to allow adequate neuropsychological testing
* Willing to undergo brain imaging
* At risk for cognitive decline, as defined by one or more of the following: Personal or family history of mood disorder, Hypothyroidism, Diabetes, Family history of Alzheimer's, APOE-4 allele

Exclusion Criteria:

* Diagnosis of possible or probable Alzheimer's disease or dementia
* Cerebrovascular disease or uncontrolled hypertension (systolic BP >170 or diastolic BP >100)
* History of myocardial infarction within previous year or unstable heart disease
* History of significant liver disease, pulmonary disease, or current cancer
* Contraindication for MRI (metal in body, claustrophobia, etc.)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women between the ages of 45 and 65 years of age, currently on estrogen therapy for 1 year prior to enrollment in study, and at risk for cognitive decline.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2003-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes in cognition and brain metabolism | Baseline and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Rasgon, MD, PhD, Principal Investigator — Stanford University School of Medicine, Dept of Psychiatry and Behavioral Sciences; Terence Ketter, MD, Principal Investigator — Stanford University; Jerome Yesavage, MD, Principal Investigator — Stanford University; Jennifer Hoblyn, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- Stanford University School of Medicine, Dept. of Psychiatry and Behavioral Sciences, Stanford, California, United States

REFERENCES:
- [Background] Rasgon NL, Small GW, Siddarth P, Miller K, Ercoli LM, Bookheimer SY, Lavretsky H, Huang SC, Barrio JR, Phelps ME. Estrogen use and brain metabolic change in older adults. A preliminary report. Psychiatry Res. 2001 Jul 1;107(1):11-8. doi: 10.1016/s0925-4927(01)00084-1. PMID 11472860
- [Background] Rasgon NL, Thomas MA, Guze BH, Fairbanks LA, Yue K, Curran JG, Rapkin AJ. Menstrual cycle-related brain metabolite changes using 1H magnetic resonance spectroscopy in premenopausal women: a pilot study. Psychiatry Res. 2001 Feb 28;106(1):47-57. doi: 10.1016/s0925-4927(00)00085-8. PMID 11231099
- [Background] Dunkin J, Rasgon N, Wagner-Steh K, David S, Altshuler L, Rapkin A. Reproductive events modify the effects of estrogen replacement therapy on cognition in healthy postmenopausal women. Psychoneuroendocrinology. 2005 Apr;30(3):284-96. doi: 10.1016/j.psyneuen.2004.09.002. PMID 15511602
- [Derived] Rasgon NL, Geist CL, Kenna HA, Wroolie TE, Williams KE, Silverman DH. Prospective randomized trial to assess effects of continuing hormone therapy on cerebral function in postmenopausal women at risk for dementia. PLoS One. 2014 Mar 12;9(3):e89095. doi: 10.1371/journal.pone.0089095. eCollection 2014. PMID 24622517